CLINICAL TRIAL: NCT02286804
Title: Evaluation of the Ulthera® System for Efficacious and Safe Treatment of Leg Telangiectasia
Brief Title: Ultherapy for the Treatment of Spider Veins on the Legs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-301
Record Dates: First submitted 2014-11-05; First posted 2014-11-10 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2015-05

CONDITIONS: Telangiectasia; Spider Veins
MeSH Terms: conditions — Telangiectasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Improvement of leg telangiectasia was determined by a masked, qualitative assessment of 2D photographs compared to baseline.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultherapy treatment (Experimental): Subjects receiving Ultherapy treatment to up to 4 spider veins
  Interventions: Device: Ultherapy

INTERVENTIONS:
Device: Ultherapy — Micro-focused ultrasound energy delivered below the surface of the skin
  Other Names: Ulthera System

SUMMARY:
Up to 30 enrolled subjects will be treated. Enrolled subjects will receive Ultherapy® treatments along each length of the spider vein. Follow-up visits will occur at 30 and 60 days post-treatment. Study images will be obtained pre-treatment, immediately post-treatment, and at each follow-up visit.

DETAILED DESCRIPTION:
This study is a prospective, single center, clinical trial to be conducted at one clinical site. Enrolled subjects will receive up to three Ultherapy® treatments at a single depth, 14 days apart, using a 10-1.5mm transducer. Treatment will be provided along each length of the spider vein and up to four veins will be treated per subject Maximum length of each vein treated is 2cm.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18 years or older.
* Subject in good health.
* Fitzpatrick Skin Types I-III.
* Understands and accepts the obligation not to undergo any other elective procedures, i.e., laser and IPL, in the areas to be treated through the follow-up period.
* Has up to 4 separate spider veins measuring up to 2 cm in length at a depth of approximately 1.0mm.
* Has lower extremity spider veins ≤1.0mm in diameter, linear or branching, and red, pink, blue and/or purple in color, as assessed by the Investigator.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the Screening Visit and be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:

  1. Postmenopausal for at least 12 months prior to study;
  2. Without a uterus and/or both ovaries; or
  3. Bilateral tubal ligation at least six months prior to study enrollment.
* Absence of physical or psychological conditions unacceptable to the investigator.
* Willingness to refrain from use of aspirin, Ibuprofen, Naproxen or any other NSAID prior to each study treatment and chronic use during the entire post-treatment study period. Washout period, if chronic user, for 4 weeks prior to the first treatment. Washout period for limited acute NSAID use, i.e., a maximum of 2-3 doses, is required in the 2 weeks prior to any study treatment visit.
* Willingness and ability to provide written consent for study-required photography and adherence to photography procedures (i.e., removal of jewelry and makeup).
* Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Presence of significant varicosities or perforator veins in the area(s) to be treated.
* Presence of large torturous varicose veins in the area(s) to be treated.
* Significant scarring in the area(s) to be treated.
* Open wounds or lesions in the area(s) to be treated.
* Active implants or metallic implants in the treatment areas.
* Presence of underlying metal hardware attached to bone from previous surgeries.
* Inability to understand the protocol or to give informed consent.
* BMI equal to or greater than 30.
* History of chronic drug or alcohol abuse.
* History of diabetes.
* History of keloid scarring, hypertrophic scarring or abnormal wound healing.
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* History of thromboembolic disease, such as deep vein thrombosis (DVT).
* History of autoimmune disease.
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
* Subjects who anticipate the need for surgery or overnight hospitalization during the study.
* Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
* Concurrent enrollment in any study involving the use of investigational devices or drugs.
* Current smoker or history of smoking in the last five years.
* History of using the following prescription medications:

  1. Accutane or other systemic retinoids within the past six months;
  2. Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix);
  3. Chronic use of non-steroidal anti-inflammatories (naproxen, ibuprofen, etc.) within the past 4 weeks;
  4. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Improvement of leg telangiectasia | 60 days post-treatment
  Determined by a masked, qualitative assessment of 2D photographs compared to baseline, based on level of clearance/improvement. Level of improvement scale:
  * 0 = 0% Improvement (None)
  * 1 = < 25% Improvement (Mild)
  * 2 = 26 to 50% Improvement (Moderate)
  * 3 = 51 to 75% Improvement (Significant)
  * 4 = 76 to 100% Improvement (Very Significant)

SECONDARY OUTCOMES:
Clinician assessment of overall aesthetic improvement | 30 days post-treatment
  Overall aesthetic improvement will be assessed using the Global Aesthetic Improvement Scale:
  1. Very Much Improved: Optimal cosmetic result in this subject.
  2. Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal for this subject.
  3. Improved: Obvious improvement in appearance from initial condition, but a re-treatment is indicated.
  4. No Change: The appearance is essentially the same as the original condition.
  5. Worse: The appearance is worse than the original condition.
Clinician assessment of overall aesthetic improvement | 60 days post-treatment
  Overall aesthetic improvement will be assessed using the Global Aesthetic Improvement Scale:
  1. Very Much Improved: Optimal cosmetic result in this subject.
  2. Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal for this subject.
  3. Improved: Obvious improvement in appearance from initial condition, but a re-treatment is indicated.
  4. No Change: The appearance is essentially the same as the original condition.
  5. Worse: The appearance is worse than the original condition.
Subject assessment of overall aesthetic improvement | 30 days post-treatment
  Overall aesthetic improvement will be assessed using the Global Aesthetic Improvement Scale:
  1. Very Much Improved: Optimal cosmetic result in this subject.
  2. Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal for this subject.
  3. Improved: Obvious improvement in appearance from initial condition, but a re-treatment is indicated.
  4. No Change: The appearance is essentially the same as the original condition.
  5. Worse: The appearance is worse than the original condition.
Subject assessment of overall aesthetic improvement | 60 days post-treatment
  Overall aesthetic improvement will be assessed using the Global Aesthetic Improvement Scale:
  1. Very Much Improved: Optimal cosmetic result in this subject.
  2. Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal for this subject.
  3. Improved: Obvious improvement in appearance from initial condition, but a re-treatment is indicated.
  4. No Change: The appearance is essentially the same as the original condition.
  5. Worse: The appearance is worse than the original condition.
Patient Satisfaction | 30 days post-treatment
  Subjects will rate their satisfaction with the outcome of their treatment based on completion of a patient satisfaction questionnaire using the following scale:
  * Very Satisfied
  * Satisfied
  * Slightly Satisfied
  * Neither Satisfied or Dissatisfied
  * Dissatisfied
Patient Satisfaction | 60 days post-treatment
  Subjects will rate their satisfaction with the outcome of their treatment based on completion of a patient satisfaction questionnaire using the following scale:
  * Very Satisfied
  * Satisfied
  * Slightly Satisfied
  * Neither Satisfied or Dissatisfied
  * Dissatisfied

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Misell, PhD, Study Director — Ulthera, Inc
Locations (1):
- Ulthera, Inc., Mesa, Arizona, United States